CLINICAL TRIAL: NCT03055650
Title: iLux Treatment for Meibomian Gland Dysfunction (MGD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tear Film Innovations, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01
Record Dates: First submitted 2017-02-10; First posted 2017-02-16 (Actual); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Evaporative Dry Eye
Keywords: Evaporative Dry Eye (EDE); Meibomian Gland Dysfunction (MGD)
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- iLux 2020 System (Experimental): Meibomian gland treatment (Day 0) according to instructions for use (IFU)/User Manual
  Interventions: Device: iLux 2020 System

INTERVENTIONS:
Device: iLux 2020 System — Medical device that applies localized heat and pressure therapy to the eyelid in order to express melted meibum from obstructed glands

SUMMARY:
The purpose of this study is to assess changes in meibomian gland function and evaporative dry eye symptoms after treatment with the iLux medical device.

DETAILED DESCRIPTION:
Alcon Research, LLC, acquired TearFilm Innovations, Inc., in December 2018. This study was designed and conducted by TearFilm Innovations, Inc. The study results were collected, analyzed, and provided by TearFilm Innovations, Inc., to Alcon Research, LLC.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older of any gender or race
2. Provision of written informed consent prior to study participation
3. Willingness and ability to return for all study visits
4. A positive history of self-reported dry eye symptoms for three months prior to the study using the Standard Patient Evaluation of Eye Dryness (SPEED) questionnaire, and a score of > 6.
5. Need for regular use of artificial tears, lubricants, or rewetting drops in both eyes
6. Evidence of meibomian gland (MG) obstruction, based on a total meibomian gland secretion score of < 12 out of a maximum score of 45, for 15 glands (5 nasal, 5 medial, 5 temporal) of the lower eyelid of each eye. Glands expressed & graded from 0 to 3 (0 = no secretion, 1 = inspissated, 2 = cloudy, 3 = clear liquid).

Exclusion Criteria:

1. History of ocular surgery including intraocular, oculo-plastic, corneal or refractive surgery within 1 year
2. Ocular trauma or herpetic keratitis within the previous 3 months
3. Cicatricial lid margin disease identified via slit lamp examination, including pemphigoid, symblepharon, etc.
4. Active ocular infection (e.g., viral, bacterial, mycobacterial, protozoan, or fungal infection of the cornea, conjunctiva, lacrimal gland, lacrimal sac, or eyelids including a hordeolum or stye)
5. Active ocular inflammation or history of chronic, recurrent ocular inflammation within prior 3 months (e.g. retinitis, macular inflammation, choroiditis, uveitis, iritis, scleritis, episcleritis, keratitis)
6. Ocular surface abnormality that may compromise corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, or map dot fingerprint dystrophy
7. Lid surface abnormalities (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis) that affect lid function in either eye
8. Anterior blepharitis (staphylococcal, demodex or seborrheic grade 3 or 4)
9. Ocular trauma, chemical burns, or limbal stem cell deficiency
10. Systemic disease conditions that cause dry eye (e.g., Stevens-Johnson syndrome, vitamin A deficiency, rheumatoid arthritis, Wegener's granulomatosis, sarcoidosis, leukemia, Riley-Day syndrome, systemic lupus erythematosus, Sjogren's syndrome)
11. Women who are pregnant, nursing, or not utilizing adequate birth control measures
12. Individuals who have either changed the dosing of systemic or ophthalmic medication within the past 30 days prior to screening or who are unable or unwilling to remain on a stable dosing regimen for the duration of the study
13. Individuals using isotretinoin (Accutane) within 1 year, cyclosporine-A (Restasis) within 2 months, or topical medications other than non-preserved artificial tears within 2 weeks.
14. Individuals using another investigational device or agent within 30 days of study participation
15. Contact lens wearers or individuals who have worn contact lenses in the last 30 days or anticipate wearing contact lenses during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2016-02-18 (Actual); Study Completion 2016-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - TearFilm Investigative Site, Encinitas, California
  - TearFilm Investigative Site, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schanzlin D, Owen JP, Klein S, Yeh TN, Merchea MM, Bullimore MA. Efficacy of the Systane iLux Thermal Pulsation System for the Treatment of Meibomian Gland Dysfunction After 1 Week and 1 Month: A Prospective Study. Eye Contact Lens. 2022 Apr 1;48(4):155-161. doi: 10.1097/ICL.0000000000000847. PMID 34620785

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 3 investigative sites located in the United States.
Pre-assignment Details: This reporting group includes all enrolled participants.
Period: Overall Study
Arm/Group | iLux 2020 System
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | iLux 2020 System
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20
  Native American | 4
  Asian | 2
  Hispanic | 2
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Meibomian Gland Secretion (MGS) Total Score
Description: Meibomian glands on the lower eyelid were assessed by the examiner using a Meibomian Gland Evaluator (MGE 1000) device while viewing the eyelid margin with a slit lamp microscope. 5 glands in 3 zones (nasal, medial, temporal) were evaluated. Each gland was scored from 0-3, for a resultant overall score of 0-45 for each eye. MGS scoring was as follows: 0 = no secretion (worst), 1 = inspissated, 2 = cloudy, 3 = clear liquid (best). A positive change value indicates an improvement. Eyes were assessed individually.
Time Frame: Baseline (Day 0 pretreatment), Week 1, Month 1
Population: All treated with available data
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | iLux 2020 System
Number analyzed (Participants) | 30
Number analyzed (eyes) | 60
score on a scale
  Change from Baseline at Week 1 | 12.3 (7.1)
  Change from Baseline at Month 1 | 14.5 (7.9)
Statistical Analysis 1: Comparison: iLux 2020 System; Change from Baseline in Meibomian Gland Secretion Total Score at Week 1; Test type: Superiority; p < 0.0001, t-test, 2 sided; Statistical significance is set at α = 0.05
Statistical Analysis 2: Comparison: iLux 2020 System; Change from Baseline in Meibomian Gland Secretion Total Score at Month 1; Test type: Superiority; p < 0.0001, t-test, 2 sided; Statistical significance is set at α = 0.05

2. Primary Outcome: Change From Baseline in Tear Break-Up Time (TBUT)
Description: The investigator instilled a drop of fluorescein into the lower eyelid and asked the patient to blink several times, then stop. The time between the last blink and the first appearance of a dark spot on the cornea (formation of a dry area) on the otherwise continuously stained tear film was recorded in seconds. 3 consecutive measurements were taken, with TBUT defined as the average of the 3 measurements. A positive change value represents A positive change value represents a more stable tear film (improvement). Eyes were assessed individually.
Time Frame: Baseline (Day 0 pretreatment), Week 1, Month 1
Population: All treated with available data
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | iLux 2020 System
Number analyzed (Participants) | 30
Number analyzed (eyes) | 60
seconds
  Change from Baseline at Week 1 | 3.6 (3.1)
  Change from Baseline at Month 1 | 4.6 (3.1)
Statistical Analysis 1: Comparison: iLux 2020 System; Change From Baseline in Tear Break-Up Time (TBUT) at Week 1; Test type: Superiority; p < 0.0001, t-test, 2 sided; Statistical significance is set at α = 0.05
Statistical Analysis 2: Comparison: iLux 2020 System; Change From Baseline in Tear Break-Up Time (TBUT) at Month 1; Test type: Superiority; p < 0.0001, t-test, 2 sided; Statistical significance is set at α = 0.05

3. Secondary Outcome: Change From Baseline in Standard Patient Evaluation of Eye Dryness (SPEED) Total Score
Description: The Standard Patient Evaluation of Eye Dryness (SPEED) survey is a validated survey that assesses both the frequency and severity of dry eye symptoms. The patient grades the frequency of symptoms (4 items) on a scale from 0 to 3 (0=never; 3=constant) and the severity of each symptom (4 items) on a scale from 0 to 4 (0=no problems; 4=intolerable). Responses to the 8 items are summed to calculate a total score ranging from 0 to 28, where 0=best and 28=worst. A negative change value indicates a perceived improvement in ocular health. Both eyes contributed to the mean.
Time Frame: Baseline (Day 0 pretreatment), Week 1, Month 1
Population: All treated with available data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iLux 2020 System
Number analyzed (Participants) | 30
score on a scale
  Change from Baseline at Week 1 | -8.6 (7.0)
  Change from Baseline at Month 1 | -9.1 (6.6)
Statistical Analysis 1: Comparison: iLux 2020 System; Change From Baseline in Standard Patient Evaluation of Eye Dryness (SPEED) Total Score at Week 1; Test type: Superiority; p < 0.0001, t-test, 2 sided; Statistical significance is set at α = 0.025
Statistical Analysis 2: Comparison: iLux 2020 System; Change From Baseline in Standard Patient Evaluation of Eye Dryness (SPEED) Total Score at Month 1; Test type: Superiority; p < 0.0001, t-test, 2 sided; Statistical significance is set at α = 0.025

4. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI) Total Score
Description: The OSDI is a validated, 12-item questionnaire used to measure ocular symptoms, visual function, and environmental factors that may affect a patient's vision. The patient grades each item on a scale from 0 to 4, where 0 is "None" and 4 is "All of the Time." Responses to the 12 items are summed, and a formula is used to calculate a total score from 0 to 100, where 0 corresponds to no disability and 100 corresponds to complete disability. A negative change value represents a perceived improvement in ocular health. Both eyes contributed to the mean.
Time Frame: Baseline (Day 0 pretreatment), Month 1
Population: All treated with available data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iLux 2020 System
Number analyzed (Participants) | 30
score on a scale | -28.5 (22.0)
Statistical Analysis 1: Comparison: iLux 2020 System; Test type: Superiority; p < 0.0001, t-test, 2 sided; Statistical significance is set at α = 0.025

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant from time of enrollment until time of study exit, approximately 4 weeks.
Description: An adverse event was defined as any untoward and unintended sign, symptom or disease temporally associated with the use of an investigational drug or device, or other protocol-imposed intervention, regardless of the suspected cause. All subjects exposed to the study treatment were evaluated for adverse events.
Groups:
- iLux 2020 System: Meibomian Gland Treatment
  iLux 2020 System: Heating and compression to express clogged meibomian glands
Arm/Group | iLux 2020 System
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes